CLINICAL TRIAL: NCT02002143
Title: Group Medical Visits (GMVs) in Primary Care: An RCT of Group-Based Versus Individual Appointments to Reduce HbA1c in Older People
Brief Title: GMVs in Primary Care: An RCT of Group-Based Versus Individual Appointments to Reduce HbA1c in Older People
Acronym: GAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government)
Responsible Party: Principal Investigator, Karim Miran-Khan, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-02812
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes; Older People; Seniors; Group Appointments; Group Medical Visits; Shared Appointments; Quality of Life; Physical Activity; Health care Utilization; Depression; Anxiety
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity; Patient Acceptance of Health Care; Depression; Anxiety Disorders | interventions — Shared Medical Appointments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Appointments (IAs) (Active Comparator): Participants randomly assigned to the "IAs" group will receive eight traditional 1-to-1 appointments, seeing their physician quarterly as per standard care in BC. They will be referred to ancillary services such as nutrition advice, counseling, and physical activity promotion according to 'usual care' practice. In addition, we will organize 4 1-hour social events for these participants annually. The 4 social events will be 1) a potluck lunch; 2) a movie night; 3) an event chosen by participants; and 4) a talent show. From our experience, these events enhance compliance to reporting and minimize dropouts. These events also serve to minimize 'socialization bias' that may otherwise potentially influence health measures including quality of life.
  Interventions: Behavioral: Individual Appointments (IAs)
- Group Appointments (GAs) (Experimental): Participants randomly assigned to the intervention group will participate in GAs of 8 patients for 1.5 hours, every 3 months for 2 years. The 3-member Care Team (MD, nurse, behaviorist) will attend each session. The nurse facilitates the session and curriculum. The MD responds to specific health questions. Patients may schedule time before or after to review their clinical results with the MD/nurse (e.g. HbAIC).
  Key elements include 1) completed pre-appt questionnaires used to identify a patient's educational needs; 2) patients use goal setting and action plans to initiate and maintain healthy behaviors; 3) each class has a designated purpose and learning objectives; 4) sessional feedback, which is used to adapt the next class (3 months later) based on patient needs.
  Interventions: Behavioral: Group Appointments

INTERVENTIONS:
Behavioral: Group Appointments — Participants randomly assigned to the intervention group will participate in GAs of 8 patients for 1.5 hours, every 3 months for 2 years. The 3-member Care Team (MD, nurse, behaviorist) will attend each session. The nurse facilitates the session and curriculum. The MD responds to specific health questions. Patients may schedule time before or after to review their clinical results with the MD/nurse (e.g. HbAIC).
  Key elements include 1) completed pre-appt questionnaires used to identify a patient's educational needs; 2) patients use goal setting and action plans to initiate and maintain healthy behaviors; 3) each class has a designated purpose and learning objectives; 4) sessional feedback, which is used to adapt the next class (3 months later) based on patient needs.
  Other Names: Shared Appointments; Group Medical Visits
  Arms: Group Appointments (GAs)
Behavioral: Individual Appointments (IAs) — Participants randomly assigned to the "IAs" group will receive eight traditional 1-to-1 appointments, seeing their physician quarterly as per standard care in BC. They will be referred to ancillary services such as nutrition advice, counseling, and physical activity promotion according to 'usual care' practice. In addition, we will organize 4 1-hour social events for these participants annually. The 4 social events will be 1) a potluck lunch; 2) a movie night; 3) an event chosen by participants; and 4) a talent show. From our experience, these events enhance compliance to reporting and minimize dropouts. These events also serve to minimize 'socialization bias' that may otherwise potentially influence health measures including quality of life.
  Arms: Individual Appointments (IAs)

SUMMARY:
Type 2 diabetes is a major problem of older people; its prevalence is greater than 20% in those aged over 65 years. Treatment such as medication, healthy nutritional choices & body weight management, as well as physical activity can reduce the impact of diabetes.

Older patients with type 2 diabetes can potentially benefit from Group Appointments, in which 8-12 patients share one appointment of about 60-120 minutes with a team of health professionals.

The team of investigators (3 people) will see the 'Group' 4 times/yr for two years. Their key measure of success will be control of glycosylated hemoglobin - HbA1C.

To address their primary and secondary research objectives the investigators will focus upon patients aged 65 years or older who have T2DM and who are being treated with oral hypoglycemic agents and diet, or diet alone.

The investigators will compare patients randomized to (A) eight Group Appointments over a 24 month period (i.e., 4 per year), led by a primary care physician [Intervention] with, (B) patients randomized to eight traditional one-to-one usual care appointments also provided by a primary care physician (Individual Appointment; [Control]). The investigators will compare (A) and (B) on selected clinical, patient-rated, and economic outcome measures.

SIGNIFICANCE: Seven Canadian provinces already have Group Appointment billing codes for physicians who lead Group Appointments. If the study's proposed health care innovation demonstrates benefits, it would be possible to 'roll out' / 'scale up' the model province- or nation-wide in Primary Care settings.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) in older people is an undisputed health problem. More than 1.1 million people diagnosed with diabetes mellitus (DM) in Canada are over the age of 65 years. Rates of T2DM in older people are accelerating even when adjusted for age. Thus, total community prevalence is increasing based on the greater number of older people, an increased rate among those older people, and improved survival rates of people with DM.

The financial burden of DM to the Canadian health care system will approach $17 billion/year by 2020. Beyond the direct health burden of T2DM, the condition is an independent risk factor for falls and dementia -two of the 'geriatric giants'. T2DM is 'an important unresolved issue previously unacknowledged' and is considered to increase 'biological age' by 2 years in those aged over 70 years.

Although treatment can improve the clinical trajectory of older people with T2DM, many do not receive guideline care. Combinations of drug treatment, physical activity, nutrition advice and body weight management, reduce risk factors, delay onset of disease and lessen the rate of complications.

Group Appointments (GAs) - also called Group Medical Visits or Shared Medical Appointments may contribute to improved T2DM care for older people in the primary care setting. The innovation in this study is to undertake research in one study to determine 1) the clinical effectiveness; 2) quality of life; and 3) economic implications of Group Appointments for older people with T2DM.

'Group Appointments' exist in various forms. Their origin is often attributed to Noffsinger and also Ward. In a Group Appointment, one physician works with a nurse and a 'behaviourist' (described on page 12c) to care for eight to twelve patients during one 60-120 minute appointment.

A recent Systematic Review of Group Appointments in T2DM performed by two current Co-Investigators (HOUSDEN, DAWES) highlighted the need for a Canadian Primary Care RCT that would extend previous research from Italy. The extension of research by this study is to have a Primary Care physician lead Group Appointments and for the RCT to include exclusively men and women aged 65 years and older.

The clinical and societal importance of T2DM in older people is not disputed. 'Diabetes mellitus is a serious condition with potentially devastating complications that affects all age groups worldwide'.

Diabetes epidemiology was reviewed in the 2013 Canadian Diabetes Practice Guidelines and Public Health Agency of Canada's 'Diabetes in Facts & Figures'. To make this literature 'critical' the investigators will focus on 1) the accelerating rate of diagnosis of type 2 diabetes in older people; 2) the challenge of delivering quality diabetes care affordably in a traditional one-to-one primary care encounter 3) the equipoise that results from international evidence for testing GAs to improve patient self-management in the absence of Canadian Primary Care research in this field; 4) a brief review of the validity and limitations of HbA1C as a measure of T2DM self-management; and 5) the theoretical framework underpinning their Group Appointment intervention.

From the 2013 Canadian Clinical Practice Guidelines for Diabetes, as of 2009, 6.8% of Canadians (2.4 million people) had the condition. This represented a 230% increase compared to prevalence estimates 11 years earlier. A decade from now, an additional 1.3 million Canadians are expected to have T2DM. Diabetes and its complications increase costs and service pressures on Canada's publicly funded healthcare system. People with diabetes were three times more likely to require hospital admission in the preceding year with longer lengths of stay.

Good metabolic control of diabetes prevents complications. This requires lifestyle and behavioural modification. In Canada, the usual clinical care for diabetes is via individual patient consultations combined with 'ad hoc' educational advice during a family practice appointment or referral to an educational support program, if available. Although traditional primary care delivery addresses clinical problems, it fails to embrace the principles of behaviour change (compliance/ adherence) that are an essential part of chronic disease management.

The Canadian Practice Guidelines for T2DM call for psychological support, exercise promotion and nutritional advice. Traditional one-to-one clinical encounters in a fee-for-service setting do not encourage such coordinated care. There is a call to improve the scope of diabetes care currently offered in Canada. The quote 'if you keep doing what you've always done, you'll keep getting what you've always got' is relevant in this setting.

Traditional one-to-one clinical encounters will always have a place in health service delivery.

However, given the common needs across patients and the burgeoning costs to treat those with T2DM - the investigators address the question, 'Is there a more effective way to encourage successful patient self-management for older people with T2DM.

Two major resources on Group Appointments relate to various medical settings (i.e., not primary care alone). The 'Bible' of Group Appointments is Dr. Edward Noffsinger's 500-page book Running Group Visits in Your Practice (2009). He describes two main types of GAs -not limited to the primary care setting. A second foundational source for Canadians in particular, is The Group Medical Appointment Manual (First Edition 2007) published by the Northern Health Authority in British Columbia (developed after a visit by Dr. Noffsinger).

In clinical trials, the most compelling data for Group Appointments providing superior control of HemoglobinAA1C come from Drs. Trento and Porta, University of Turin, Italy. Patients who attended structured Group Appointments decreased their HbA1C by 0.9% (Effect size 0.56) compared with control group counterparts. There are a number of differences between these studies and what the investigators propose. First, studies in Turin and around Italy took place in 'hospital-based clinics', not regular primary care settings. Second, participants in the Turin studies were 64years, on average -younger than in our proposed study. Third, Turin studies did not include a generic quality of life measure (e.g. EQ-5D) and did not estimate health utilities. Fourth, health economic implications cannot be extrapolated from the Italian to the Canadian health system.

Considering all published RCTs, HOUSDEN and DAWES (co-investigators) found a significant 0.46% reduction in HbA1C across 10 RCTs that met their inclusion criteria. However, in a 12- month US Veteran Affairs Medical Centre trial, GA patients had only a 0.3% improvement over patients randomized to individual care (effect size 0.21). Other than study duration, the approach between the US and University of Turin studies appeared similar.

The aforementioned HOUSDEN and DAWES' systematic review highlighted that no RCT in the Primary Care setting examined Group Appointments as a vehicle to improve patient management as measured by HbAIC or another clinical measure. Previous published papers describing T2DM Group Appointments in the Primary Care setting focused on patient satisfaction and physician perception.

Such research provides valuable insight into barriers and facilitators to Group Appointments. However, no studies answered the question 'Do Primary Care-led Group Appointments improve metabolic control in diabetes?' HOUSDEN reported that duration of Group Appointments (i.e., 24-months) was significantly associated with outcome (approximately 0.25% lower HbA1C per year) but number of GAs was not. That informed the decision of the investigators to conduct an RCT across two years.

The rationale for Group Appointments builds on the social cognitive theory and transtheoretical stages of change at the individual level and brings to bear group dynamics that are unavailable in an Individual Appointment. The investigators emphasize that GAs combine three elements: 1) medical care; 2) disease-specific education (e.g. the significance of HbA1C, healthy food choices); and 3) life skills development such as goal setting, action planning, and problem-solving.

Patients who attend the Group Appointments are, by definition, in the 'post-intentional' phase (transtheoretical model) when they receive education. They know their diagnosis and recognize the need to do something about it. Thus, Group Appointments move beyond mere education of medical facts and are 'dynamic' in that the curriculum will focus on key challenges that surface in the process of turning goals into action.

Collectively, these components will help patients adopt healthier lifestyles (action) and also maintain these health behavior changes when they experience setbacks or failures (coping). This is consistent with the transtheoretical model and well as the health action process approach.

Note that the Group Appointments also reinforce self-efficacy and emotional support.

This contrasts with a traditional primary care individual appointment where 1) the clinician may or may not make time for counseling in a busy schedule or 2) gives generic verbal advice or referral without attention to specific nutrition or physical activity goals that may be most appropriate for the patient. The investigators propose elements for GAs that are consistent with best evidence and patient preference.

On the one hand, Group Appointments may at first seem a logical component of the diabetes continuum of care. A proportion of primary care practices, including those of our collaborators offer them. There is Provincial Government and British Columbia (BC) Medical Association (BCMA) (through the General Practice Services Committee) endorsement. Yet there remain no quantitative metabolic (HbA1C) or economic data (QALY/health care utilization) on the outcomes of Group Appointments specifically for elderly patients with T2DM in the Canadian Primary Care setting.

Therefore, this rigorous review of the literature suggests - there is as yet NO clear Canadian evidence that would convince policymakers to invest in Primary care-led Group Appointment for older people with T2DM unless further evidence was obtained to show they work. The investigators propose to address this gap. They will conduct measurements at 0 (baseline), 12 (mid-intervention) and 24 (end of-intervention), months. The investigators assess primary outcomes at 24 months but will follow-up to evaluate change at 36 months (12-month follow-up). In addition, the investigators will obtain three-monthly data for blood tests as part of routine patient management before each of the three-monthly Group Appointments (Intervention) and at individual patient appointments (usual care). At these three-monthly intervals a research assistant (RA#1) will administer the Health Resource Utilization (HUI3) collection instrument and the EQ-5D.

SIGNIFICANCE: Despite the clinical burden of T2DM among older Canadians, and the potential for the primary care system to deliver innovative multidisciplinary care and education, there have been no randomized controlled trials (RCTs) with that goal. The "GAP" study will apply conceptual clinical innovations in Group Appointments in the primary care setting to the health need of older adults with diabetes. There is a need for quantitative Canadian research in GAs broadly and the investigators target the substantial clinical problem - diabetes in older people. Do primary care led, Group Appointments reduce HbA1C, improve quality of life and do so at a reasonable price? If the answer is encouraging, there is potential to 'scale-up' the model via divisions, provinces and ultimately nationwide.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years old;
* have at least a 12-month history of T2DM based on the Canadian Diabetes Guidelines;
* be community-dwelling;
* live within 30km of their GP clinic in Abbotsford, BC (Canada);
* able to comply with scheduled visits, treatment plan, and other trial procedures;
* read, write, and speak English;
* acceptable auditory acuity to participate in the Group Appointments and visual acuity to participate in the research;
* provide a personally signed and dated informed consent;
* able to walk independently;
* Inclusion will be based on medical history, vital signs, physical examination by study physicians, and written recommendation by family physician, indicating the patient's appropriateness to participate.

Exclusion Criteria:

* using insulin to treat diabetes to increase the homogeneity of the sample;
* at high risk for cardiac complications during exercise and/or unable to self-regulate activity or to understand recommended activity level (i.e., Class C of the American Heart Risk Stratification Criteria);
* Mini-Mental State Examination (MMSE)[51] score of ≤ 24 at screening;
* have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility;
* taking medications that may negatively affect the ability to undertake a simple walking program safely (e.g. beta blockers);
* planning to participate, or already enrolled in, a clinical drug trial concurrent to this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Patients' control (decreased levels) of HemoglobinA1C (clinical) | Changes from baseline at 24 months
  The investigators will measure Hemoglobin A1C (%, primary outcome), utilizing the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.

SECONDARY OUTCOMES:
Resting systolic blood pressure (mmHg)) (clinical) | Changes from baseline at 12 months
  The investigators will assess resting systolic blood pressure with an automated BP device BPTRU™.
Resting systolic blood pressure (mmHg)) (clinical) | Changes from baseline at 24 months
  The investigators will assess resting systolic blood pressure with an automated BP device BPTRU™.
Resting systolic blood pressure (mmHg)) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess resting systolic blood pressure with an automated BP device BPTRU™.
Resting diastolic blood pressure (mmHg)) (clinical) | Changes from baseline at 12 months
  The investigators will assess resting diastolic blood pressure with an automated BP device BPTRU™.
Resting diastolic blood pressure (mmHg)) (clinical) | Changes from baseline at 24 months
  The investigators will assess resting diastolic blood pressure with an automated BP device BPTRU™.
Resting diastolic blood pressure (mmHg)) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess resting diastolic blood pressure with an automated BP device BPTRU™.
Electrical activity of the heart (ECG) (clinical) | Changes from baseline at 12 months
  The investigators will assess cardiovascular disease risk factors by 12-lead ECG (10 minutes).
Electrical activity of the heart (ECG) (clinical) | Changes from baseline at 24 months
  The investigators will assess cardiovascular disease risk factors by 12-lead ECG (10 minutes).
Electrical activity of the heart (ECG) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess cardiovascular disease risk factors by 12-lead ECG (10 minutes).
C-reactive protein (mg/L) (clinical) | Changes from baseline at 12 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
C-reactive protein (mg/L) (clinical) | Changes from baseline at 24 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
C-reactive protein (mg/L) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
plasma glucose (mmol/L) (clinical) | Changes from baseline at 12 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
plasma glucose (mmol/L) (clinical) | Changes from baseline at 24 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
plasma glucose (mmol/L) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
High-density lipoprotein - cholesterol (HDL-C; mmol/L) (clinical) | Changes from baseline at 12 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
High-density lipoprotein - cholesterol (HDL-C; mmol/L) (clinical) | Changes from baseline at 24 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
High-density lipoprotein - cholesterol (HDL-C; mmol/L) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Fasting low-density lipoprotein (LDL; mmol/L) (clinical) | Changes from baseline at 12 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Fasting low-density lipoprotein (LDL; mmol/L) (clinical) | Changes from baseline at 24 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Fasting low-density lipoprotein (LDL; mmol/L) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Triglycerides (mmol/L) (clinical) | Changes from baseline at 12 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Triglycerides (mmol/L) (clinical) | Changes from baseline at 24 months
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Triglycerides (mmol/L) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will utilize the phlebotomy unit in the CHHM Mobile Lab to collect a non-fasting blood sample (standard techniques). They will request that study participants not engage in any physical activity, or consume alcohol/caffeine 24 hours prior to measurement. Collected samples will be refrigerated in the Mobile Lab and transported the same day to the Vancouver General Hospital Pathology Lab for analysis as per current standard methods.
Height (cm), weight (kg), waist & hip circumference (cm), fat and muscle mass (g) (clinical) | Changes from baseline at 12 months
  Height (cm): The investigators will use the wall-mounted stadiometer (Rosscraft Inc). Weight (kg): Participants remove shoes and stand on an electronic scale (Seca Model 242, Hanover, MD). For height and weight, duplicate measures are taken unless measures differ by ±0.4 cm or ±0.2 kg, when a third measure is taken. The investigators will calculate body mass index (BMI) as wt/ht2. Waist circumference (cm): The investigators use a flexible steel tape. In older adults, it is most convenient to measure at the umbilical level. The investigators obtain two measures during minimal respiration and record to the nearest 0.1 cm. They perform a third measure if the difference between the first two measures is greater than 0.2 cm. The investigators use the mean of two and the median of three measurements for analysis for all measures. Fat and muscle mass (g): The investigators will assess total body fat mass (g) and muscle mass (g) by DXA (Hologic QDR 4500W,Hologic Inc., Waltham, MA).
Height (cm), weight (kg), waist & hip circumference (cm), fat and muscle mass (g) (clinical) | Changes from baseline at 24 months
  Height (cm): The investigators will use the wall-mounted stadiometer (Rosscraft Inc). Weight (kg): Participants remove shoes and stand on an electronic scale (Seca Model 242, Hanover, MD). For height and weight, duplicate measures are taken unless measures differ by ±0.4 cm or ±0.2 kg, when a third measure is taken. The investigators will calculate body mass index (BMI) as wt/ht2. Waist circumference (cm): The investigators use a flexible steel tape. In older adults, it is most convenient to measure at the umbilical level. The investigators obtain two measures during minimal respiration and record to the nearest 0.1 cm. They perform a third measure if the difference between the first two measures is greater than 0.2 cm. The investigators use the mean of two and the median of three measurements for analysis for all measures. Fat and muscle mass (g): The investigators will assess total body fat mass (g) and muscle mass (g) by DXA (Hologic QDR 4500W,Hologic Inc., Waltham, MA).
Height (cm), weight (kg), waist & hip circumference (cm), fat and muscle mass (g) (clinical) | Changes from baseline at 36 months (1-year post-intervention)
  Height (cm): The investigators will use the wall-mounted stadiometer (Rosscraft Inc). Weight (kg): Participants remove shoes and stand on an electronic scale (Seca Model 242, Hanover, MD). For height and weight, duplicate measures are taken unless measures differ by ±0.4 cm or ±0.2 kg, when a third measure is taken. The investigators will calculate body mass index (BMI) as wt/ht2. Waist circumference (cm): The investigators use a flexible steel tape. In older adults, it is most convenient to measure at the umbilical level. The investigators obtain two measures during minimal respiration and record to the nearest 0.1 cm. They perform a third measure if the difference between the first two measures is greater than 0.2 cm. The investigators use the mean of two and the median of three measurements for analysis for all measures. Fat and muscle mass (g): The investigators will assess total body fat mass (g) and muscle mass (g) by DXA (Hologic QDR 4500W,Hologic Inc., Waltham, MA).
Quality of life (as measured by the health state utility values of EQ-5D3L questionnaire (patient-reported quality of life/economic)) | Changes from baseline at 12 months
  QALYs are calculated based on the quality of life of a patient (measured using health utilities) in a given health state and the time spent in that health state. The EQ-5D enables QALYs to be estimated. This captures the gains from reduced morbidity and reduced mortality by assigning quality weights at specific time points to an intervention that are based on preferences, anchored on perfect health and death, and measured on an interval scale. Economic analyses will be conducted from the BC Ministry of Health perspective and will capture the time horizon of the trial (24 months).
Quality of life (as measured by the health state utility values of EQ-5D3L questionnaire (patient-reported quality of life/economic)) | Changes from baseline at 24 months
  QALYs are calculated based on the quality of life of a patient (measured using health utilities) in a given health state and the time spent in that health state. The EQ-5D enables QALYs to be estimated. This captures the gains from reduced morbidity and reduced mortality by assigning quality weights at specific time points to an intervention that are based on preferences, anchored on perfect health and death, and measured on an interval scale. Economic analyses will be conducted from the BC Ministry of Health perspective and will capture the time horizon of the trial (24 months).
Quality of life (as measured by the health state utility values of EQ-5D3L questionnaire (patient-reported quality of life/economic)) | Changes from baseline at 36 months (1-year post-intervention)
  QALYs are calculated based on the quality of life of a patient (measured using health utilities) in a given health state and the time spent in that health state. The EQ-5D enables QALYs to be estimated. This captures the gains from reduced morbidity and reduced mortality by assigning quality weights at specific time points to an intervention that are based on preferences, anchored on perfect health and death, and measured on an interval scale. Economic analyses will be conducted from the BC Ministry of Health perspective and will capture the time horizon of the trial (24 months).
Health Care Utilization | Changes from baseline at 12 months
  The investigators' economic evaluation will examine the incremental costs and benefits generated by using the Group Medical Appointments intervention versus usual care. The outcome of their cost utility analysis is the incremental cost effectiveness ratio (ICER).
  By definition, an ICER is the difference between the mean costs of providing the competing interventions divided by the difference in effectiveness (i.e., QALYs), where the ICER = Δ Cost / Δ Effect. Dr. Marra will conduct a prospective economic evaluation alongside the clinical trial to 1) estimate the mean/participant and total health care resource utilization and costs associated with Group Appointments and usual care; 2) determine the QoL as measured by health state utility values; and 3) conduct a cost-utility analysis. The cost-utility analysis will be assessed in terms of incremental cost per quality adjusted life year (QALY).
  Our instruments are the EQ-5D-3L and Heath Resource Utilization (HRU) questionnaires.
Health Care Utilization | Changes from baseline at 24 months
  The investigators' economic evaluation will examine the incremental costs and benefits generated by using the Group Medical Appointments intervention versus usual care. The outcome of their cost utility analysis is the incremental cost effectiveness ratio (ICER).
  By definition, an ICER is the difference between the mean costs of providing the competing interventions divided by the difference in effectiveness (i.e., QALYs), where the ICER = Δ Cost / Δ Effect. Dr. Marra will conduct a prospective economic evaluation alongside the clinical trial to 1) estimate the mean/participant and total health care resource utilization and costs associated with Group Appointments and usual care; 2) determine the QoL as measured by health state utility values; and 3) conduct a cost-utility analysis. The cost-utility analysis will be assessed in terms of incremental cost per quality adjusted life year (QALY).
  Our instruments are the EQ-5D-3L and Heath Resource Utilization (HRU) questionnaires.
Health Care Utilization | Changes from baseline at 36 months (1-year post-intervention)
  The investigators' economic evaluation will examine the incremental costs and benefits generated by using the Group Medical Appointments intervention versus usual care. The outcome of their cost utility analysis is the incremental cost effectiveness ratio (ICER).
  By definition, an ICER is the difference between the mean costs of providing the competing interventions divided by the difference in effectiveness (i.e., QALYs), where the ICER = Δ Cost / Δ Effect. Dr. Marra will conduct a prospective economic evaluation alongside the clinical trial to 1) estimate the mean/participant and total health care resource utilization and costs associated with Group Appointments and usual care; 2) determine the QoL as measured by health state utility values; and 3) conduct a cost-utility analysis. The cost-utility analysis will be assessed in terms of incremental cost per quality adjusted life year (QALY).
  Our instruments are the EQ-5D-3L and Heath Resource Utilization (HRU) questionnaires.
Anxiety | Changes from baseline at 12 months
  The investigators will assess anxiety with the recommended Generalized Anxiety Disorder 7-item (GAD-7) scale. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for generalised anxiety disorder. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%), and post-traumatic stress disorder (sensitivity 66%, specificity 81%).
  The GAD-7 offer clinicians concise, self-administered screening and diagnostic tools for mental health disorders.
Anxiety | Changes from baseline at 24 months
  The investigators will assess anxiety with the recommended Generalized Anxiety Disorder 7-item (GAD-7) scale. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for generalised anxiety disorder. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%), and post-traumatic stress disorder (sensitivity 66%, specificity 81%).
  The GAD-7 offer clinicians concise, self-administered screening and diagnostic tools for mental health disorders.
Anxiety | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess anxiety with the recommended Generalized Anxiety Disorder 7-item (GAD-7) scale. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for generalised anxiety disorder. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%), and post-traumatic stress disorder (sensitivity 66%, specificity 81%).
  The GAD-7 offer clinicians concise, self-administered screening and diagnostic tools for mental health disorders.
Depression | Changes from baseline at 12 months
  The investigators will assess depression with the recommended Geriatric Depression Scale (GDS). The GDS is a 30-item self-report assessment used to identify depression in the elderly. The scale was first developed in 1982 by J.A. Yesavage and others.
Depression | Changes from baseline at 24 months
  The investigators will assess depression with the recommended Geriatric Depression Scale (GDS). The GDS is a 30-item self-report assessment used to identify depression in the elderly. The scale was first developed in 1982 by J.A. Yesavage and others.
Depression | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess depression with the recommended Geriatric Depression Scale (GDS). The GDS is a 30-item self-report assessment used to identify depression in the elderly. The scale was first developed in 1982 by J.A. Yesavage and others.
Satisfaction With Life Scale | Changes from baseline at 12 months
  The Satisfaction With Life Scale (SWLS) is a measure of life satisfaction developed by Ed Diener and colleagues (Diener, Emmons, Larsen & Griffin, 1985). The SWLS consists of 5-items that are completed by the individual whose life satisfaction is being measured.
Satisfaction With Life Scale | Changes from baseline at 24 months
  The Satisfaction With Life Scale (SWLS) is a measure of life satisfaction developed by Ed Diener and colleagues (Diener, Emmons, Larsen & Griffin, 1985). The SWLS consists of 5-items that are completed by the individual whose life satisfaction is being measured.
Satisfaction With Life Scale | Changes from baseline at 36 months (1-year post-intervention)
  The Satisfaction With Life Scale (SWLS) is a measure of life satisfaction developed by Ed Diener and colleagues (Diener, Emmons, Larsen & Griffin, 1985). The SWLS consists of 5-items that are completed by the individual whose life satisfaction is being measured.
Physical Activity (PASE) | Changes from baseline at 12 months
  The investigators will assess physical activity with the valid and reliable Physical Activities Scale for the Elderly (PASE) questionnaire. PASE was designed for those aged 65 years and older; participants use a 12-item scale to self-report the hours per day (average) spent participating in leisure, household, and occupational physical activities over the previous seven-day period. Physical activity is an important covariate in this study.
Physical Activity (PASE) | Changes from baseline at 24 months
  The investigators will assess physical activity with the valid and reliable Physical Activities Scale for the Elderly (PASE) questionnaire. PASE was designed for those aged 65 years and older; participants use a 12-item scale to self-report the hours per day (average) spent participating in leisure, household, and occupational physical activities over the previous seven-day period. Physical activity is an important covariate in this study.
Physical Activity (PASE) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess physical activity with the valid and reliable Physical Activities Scale for the Elderly (PASE) questionnaire. PASE was designed for those aged 65 years and older; participants use a 12-item scale to self-report the hours per day (average) spent participating in leisure, household, and occupational physical activities over the previous seven-day period. Physical activity is an important covariate in this study.
Physical Activity (SenseWear) | Changes from baseline at 12 months
  The investigators will assess physical activity with the valid and reliable SenseWear armband, measuring steps/per day, energy expenditure (calories), and hours of activity (METs (sedentary, moderate, vigorous, very vigorous)). Participants will wear the armband for seven consecutive days, including while sleeping.
Physical Activity (SenseWear) | Changes from baseline at 24 months
  The investigators will assess physical activity with the valid and reliable SenseWear armband, measuring steps/per day, energy expenditure (calories), and hours of activity (METs (sedentary, moderate, vigorous, very vigorous)). Participants will wear the armband for seven consecutive days, including while sleeping.
Physical Activity (SenseWear) | Changes from baseline at 36 months (1-year post-intervention)
  The investigators will assess physical activity with the valid and reliable SenseWear armband, measuring steps/per day, energy expenditure (calories), and hours of activity (METs (sedentary, moderate, vigorous, very vigorous)). Participants will wear the armband for seven consecutive days, including while sleeping.
Goal Setting and Action Planning | Baseline
  Behavioural principles underpinning the intervention: Assistant Professor and Canada Research Chair HOPPMANN leads the behavioural aspects of the study. From her experience in psychological aging research and everyday health behaviours she designs Group Appointments to help patients 1) set realistic health goals; 2) identify good opportunities to translate those health goals into action (action planning); and 3) proactively map out strategies that maintain health behaviours in the face of challenges (coping planning).
  The investigators will utilize a psychology / goal setting questionnaire.
Goal Setting and Action Planning | Changes from baseline at 12 months
  Behavioural principles underpinning the intervention: Assistant Professor and Canada Research Chair HOPPMANN leads the behavioural aspects of the study. From her experience in psychological aging research and everyday health behaviours she designs Group Appointments to help patients 1) set realistic health goals; 2) identify good opportunities to translate those health goals into action (action planning); and 3) proactively map out strategies that maintain health behaviours in the face of challenges (coping planning).
  The investigators will utilize a psychology / goal setting questionnaire.
Goal Setting and Action Planning | Changes from baseline at 24 months
  Behavioural principles underpinning the intervention: Assistant Professor and Canada Research Chair HOPPMANN leads the behavioural aspects of the study. From her experience in psychological aging research and everyday health behaviours she designs Group Appointments to help patients 1) set realistic health goals; 2) identify good opportunities to translate those health goals into action (action planning); and 3) proactively map out strategies that maintain health behaviours in the face of challenges (coping planning).
  The investigators will utilize a psychology / goal setting questionnaire.
Goal Setting and Action Planning | Changes from baseline at 36 months
  Behavioural principles underpinning the intervention: Assistant Professor and Canada Research Chair HOPPMANN leads the behavioural aspects of the study. From her experience in psychological aging research and everyday health behaviours she designs Group Appointments to help patients 1) set realistic health goals; 2) identify good opportunities to translate those health goals into action (action planning); and 3) proactively map out strategies that maintain health behaviours in the face of challenges (coping planning).
  The investigators will utilize a psychology / goal setting questionnaire.
Food Diary | Baseline
  Investigators will assess nutritional intake, using a three-day food diary.
Food Diary | Changes from baseline at 12 months
  Investigators will assess nutritional intake, using a three-day food diary.
Food Diary | Changes from baseline at 24 months
  Investigators will assess nutritional intake, using a three-day food diary.
Food Diary | Changes from baseline at 36 months (1-year post-intervention)
  Investigators will assess nutritional intake, using a three-day food diary.
Patient Self-Management | Baseline
  Investigators will assess patient self-management, using the Patient Activation Measure (PAM) questionnaire. Patient self-management has been identified as a key component to the management of T2DM (CDA/ADA Practice Guidelines). Patients who have the skills, ability, and willingness to manage their own health have better health outcomes. The PAM questionnaire has been tested extensively across a number of different languages, cultures, and demographic groups, and among people with different health conditions.
Patient Self-Management | Changes from baseline at 12 months
  Investigators will assess patient self-management, using the Patient Activation Measure (PAM) questionnaire. Patient self-management has been identified as a key component to the management of T2DM (CDA/ADA Practice Guidelines). Patients who have the skills, ability, and willingness to manage their own health have better health outcomes. The PAM questionnaire has been tested extensively across a number of different languages, cultures, and demographic groups, and among people with different health conditions.
Patient Self-Management | Changes from baseline at 24 months
  Investigators will assess patient self-management, using the Patient Activation Measure (PAM) questionnaire. Patient self-management has been identified as a key component to the management of T2DM (CDA/ADA Practice Guidelines). Patients who have the skills, ability, and willingness to manage their own health have better health outcomes. The PAM questionnaire has been tested extensively across a number of different languages, cultures, and demographic groups, and among people with different health conditions.
Patient Self-Management | Changes from baseline at 36 months (1-year post-intervention)
  Investigators will assess patient self-management, using the Patient Activation Measure (PAM) questionnaire. Patient self-management has been identified as a key component to the management of T2DM (CDA/ADA Practice Guidelines). Patients who have the skills, ability, and willingness to manage their own health have better health outcomes. The PAM questionnaire has been tested extensively across a number of different languages, cultures, and demographic groups, and among people with different health conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Miran-Khan, MD, PhD, MBA, Principal Investigator — Centre for Hip Health and Mobility (University of British Columbia); Jennifer Davis, PhD, Study Director — UBC Department of Population & Public Health; Martin Dawes, MB.BS, MD, Study Director — UBC Department of Family Practice; Christiane Hoppmann, PhD, Study Director — UBC Psychology Department; Teresa Liu-Ambrose, PhD, PT, Study Director — UBC Department of Physical Therapy; Ken Madden, MD, Study Director — UBC Department of Medicine (Geriatric Medicine); Carlo Marra, Pharm.D, PhD, Study Director — UBC Faculty of Pharmaceutical Sciences; Adriaan Windt, MD, Study Director — UBC Department of Family Practice; Laura Housden, MN-NP(F), Study Director — UBC School of Nursing
Locations (2):
- Canada (2):
  - Gateway Clinic / Kent Place Clinic, Abbotsford, British Columbia
  - Centre for Hip Health and Mobility (Vancouver Coastal Health Research Institute/University of British Columbia), Vancouver, British Columbia

REFERENCES:
- [Background] Public Health Agency of Canada. Diabetes in Canada: Facts and figures from a public health perspective 2011. Ottawa: Government of Canada, 2011.
- [Background] Lysy Z, Booth GL, Shah BR, Austin PC, Luo J, Lipscombe LL. The impact of income on the incidence of diabetes: a population-based study. Diabetes Res Clin Pract. 2013 Mar;99(3):372-9. doi: 10.1016/j.diabres.2012.12.005. Epub 2013 Jan 8. PMID 23305902
- [Background] Dyck R, Karunanayake C, Pahwa P, Hagel L, Lawson J, Rennie D, Dosman J; Saskatchewan Rural Health Study Group. Prevalence, risk factors and co-morbidities of diabetes among adults in rural Saskatchewan: the influence of farm residence and agriculture-related exposures. BMC Public Health. 2013 Jan 5;13:7. doi: 10.1186/1471-2458-13-7. PMID 23289729
- [Background] Cauch-Dudek K, Victor JC, Sigmond M, Shah BR. Disparities in attendance at diabetes self-management education programs after diagnosis in Ontario, Canada: a cohort study. BMC Public Health. 2013 Jan 30;13:85. doi: 10.1186/1471-2458-13-85. PMID 23360373
- [Background] Meneilly GS. Diabetes in the elderly. Med Clin North Am. 2006 Sep;90(5):909-23. doi: 10.1016/j.mcna.2006.05.011. PMID 16962849
- [Background] Doucet G, Beatty M. The cost of diabetes in Canada: the economic Tsunami. Can J Diabetes 2010;34:27-29
- [Background] Caro JJ, Getsios D, Caro I, Klittich WS, O'Brien JA. Economic evaluation of therapeutic interventions to prevent Type 2 diabetes in Canada. Diabet Med. 2004 Nov;21(11):1229-36. doi: 10.1111/j.1464-5491.2004.01330.x. PMID 15498090
- [Background] Moffatt E, Shack LG, Petz GJ, Sauve JK, Hayward K, Colman R. The cost of obesity and overweight in 2005: a case study of Alberta, Canada. Can J Public Health. 2011 Mar-Apr;102(2):144-8. doi: 10.1007/BF03404164. PMID 21608388
- [Background] Volpato S, Leveille SG, Blaum C, Fried LP, Guralnik JM. Risk factors for falls in older disabled women with diabetes: the women's health and aging study. J Gerontol A Biol Sci Med Sci. 2005 Dec;60(12):1539-45. doi: 10.1093/gerona/60.12.1539. PMID 16424285
- [Background] Crane PK, Walker R, Larson EB. Glucose levels and risk of dementia. N Engl J Med. 2013 Nov 7;369(19):1863-4. doi: 10.1056/NEJMc1311765. No abstract available. PMID 24195563
- [Background] Lam R, Gallinaro A, Adleman J. Medical Problems Referred to a Care of the Elderly Physician: Insight for Future Geriatrics CME. Can Geriatr J. 2013 Sep 4;16(3):114-9. doi: 10.5770/cgj.16.58. eCollection 2013. PMID 23983827
- [Background] Hubbard RE, Andrew MK, Fallah N, Rockwood K. Comparison of the prognostic importance of diagnosed diabetes, co-morbidity and frailty in older people. Diabet Med. 2010 May;27(5):603-6. doi: 10.1111/j.1464-5491.2010.02977.x. PMID 20536960
- [Background] Alexander GC, Sehgal NL, Moloney RM, Stafford RS. National trends in treatment of type 2 diabetes mellitus, 1994-2007. Arch Intern Med. 2008 Oct 27;168(19):2088-94. doi: 10.1001/archinte.168.19.2088. PMID 18955637
- [Background] Furler J, Hii JW, Liew D, Blackberry I, Best J, Segal L, Young D. The "cost" of treating to target: cross-sectional analysis of patients with poorly controlled type 2 diabetes in Australian general practice. BMC Fam Pract. 2013 Mar 8;14:32. doi: 10.1186/1471-2296-14-32. PMID 23510207
- [Background] Teoh H, Despres JP, Dufour R, Fitchett DH, Goldin L, Goodman SG, Harris SB, Langer A, Lau DC, Lonn EM, John Mancini GB, McFarlane PA, Poirier P, Rabasa-Lhoret R, Tan MK, Leiter LA. Identification and management of patients at elevated cardiometabolic risk in canadian primary care: how well are we doing? Can J Cardiol. 2013 Aug;29(8):960-8. doi: 10.1016/j.cjca.2012.12.001. Epub 2013 Mar 7. PMID 23465284
- [Background] Umpierre D, Ribeiro PA, Schaan BD, Ribeiro JP. Volume of supervised exercise training impacts glycaemic control in patients with type 2 diabetes: a systematic review with meta-regression analysis. Diabetologia. 2013 Feb;56(2):242-51. doi: 10.1007/s00125-012-2774-z. Epub 2012 Nov 16. PMID 23160642
- [Background] Ferchak CV, Meneghini LF. Obesity, bariatric surgery and type 2 diabetes--a systematic review. Diabetes Metab Res Rev. 2004 Nov-Dec;20(6):438-45. doi: 10.1002/dmrr.507. PMID 15386803
- [Background] Staimez LR, Weber MB, Narayan KM, Oza-Frank R. A systematic review of overweight, obesity, and type 2 diabetes among Asian American subgroups. Curr Diabetes Rev. 2013 Jul;9(4):312-31. doi: 10.2174/15733998113099990061. PMID 23590534
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Knowler WC. Prevention of type 2 diabetes: comment on "Lifestyle modification and prevention of type 2 diabetes in overweight Japanese with impaired fasting glucose levels". Arch Intern Med. 2011 Aug 8;171(15):1361-2. doi: 10.1001/archinternmed.2011.367. No abstract available. PMID 21824949
- [Background] Buehler AM, Cavalcanti AB, Berwanger O, Figueiro M, Laranjeira LN, Zazula AD, Kioshi B, Bugano DG, Santucci E, Sbruzzi G, Guimaraes HP, Carvalho VO, Bordin SA. Effect of tight blood glucose control versus conventional control in patients with type 2 diabetes mellitus: a systematic review with meta-analysis of randomized controlled trials. Cardiovasc Ther. 2013 Jun;31(3):147-60. doi: 10.1111/j.1755-5922.2011.00308.x. Epub 2011 Dec 29. PMID 22212499
- [Background] Al Sayah F, Williams B, Johnson JA. Measuring health literacy in individuals with diabetes: a systematic review and evaluation of available measures. Health Educ Behav. 2013 Feb;40(1):42-55. doi: 10.1177/1090198111436341. Epub 2012 Apr 9. PMID 22491040
- [Background] Noffsinger E. Running Group Visits in Your Practice. NY, New York: Springer, 2009.
- [Background] Northern Health Authority. The Group Medical Appointment Manual First Edition 2007: Northern Health Authority 2007.
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Goossens ME, Rutten-van Molken MP, Vlaeyen JW, van der Linden SM. The cost diary: a method to measure direct and indirect costs in cost-effectiveness research. J Clin Epidemiol. 2000 Jul;53(7):688-95. doi: 10.1016/s0895-4356(99)00177-8. PMID 10941945
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Booth G, Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Methods. Can J Diabetes. 2013 Apr;37 Suppl 1:S4-7. doi: 10.1016/j.jcjd.2013.01.010. Epub 2013 Mar 26. No abstract available. PMID 24070961
- [Background] Manns B, Hemmelgarn B, Tonelli M, Au F, Chiasson TC, Dong J, Klarenbach S; Alberta Kidney Disease Network. Population based screening for chronic kidney disease: cost effectiveness study. BMJ. 2010 Nov 8;341:c5869. doi: 10.1136/bmj.c5869. PMID 21059726
- [Background] Rein DB, Wittenborn JS, Zhang X, Allaire BA, Song MS, Klein R, Saaddine JB; Vision Cost-Effectiveness Study Group. The cost-effectiveness of three screening alternatives for people with diabetes with no or early diabetic retinopathy. Health Serv Res. 2011 Oct;46(5):1534-61. doi: 10.1111/j.1475-6773.2011.01263.x. Epub 2011 Apr 14. PMID 21492158
- [Background] Steinsbekk A, Rygg LO, Lisulo M, Rise MB, Fretheim A. Group based diabetes self-management education compared to routine treatment for people with type 2 diabetes mellitus. A systematic review with meta-analysis. BMC Health Serv Res. 2012 Jul 23;12:213. doi: 10.1186/1472-6963-12-213. PMID 22824531
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Trento M, Passera P, Tomalino M, Bajardi M, Pomero F, Allione A, Vaccari P, Molinatti GM, Porta M. Group visits improve metabolic control in type 2 diabetes: a 2-year follow-up. Diabetes Care. 2001 Jun;24(6):995-1000. doi: 10.2337/diacare.24.6.995. PMID 11375359
- [Background] Trento M, Gamba S, Gentile L, Grassi G, Miselli V, Morone G, Passera P, Tonutti L, Tomalino M, Bondonio P, Cavallo F, Porta M; ROMEO Investigators. Rethink Organization to iMprove Education and Outcomes (ROMEO): a multicenter randomized trial of lifestyle intervention by group care to manage type 2 diabetes. Diabetes Care. 2010 Apr;33(4):745-7. doi: 10.2337/dc09-2024. Epub 2010 Jan 26. PMID 20103547
- [Background] Housden L, Wong ST, Dawes M. Effectiveness of group medical visits for improving diabetes care: a systematic review and meta-analysis. CMAJ. 2013 Sep 17;185(13):E635-44. doi: 10.1503/cmaj.130053. Epub 2013 Aug 12. PMID 23939218
- [Background] Edelman D, Fredrickson SK, Melnyk SD, Coffman CJ, Jeffreys AS, Datta S, Jackson GL, Harris AC, Hamilton NS, Stewart H, Stein J, Weinberger M. Medical clinics versus usual care for patients with both diabetes and hypertension: a randomized trial. Ann Intern Med. 2010 Jun 1;152(11):689-96. doi: 10.7326/0003-4819-152-11-201006010-00001. PMID 20513826
- [Background] Lavoie JG, Wong ST, Chongo M, Browne AJ, MacLeod ML, Ulrich C. Group medical visits can deliver on patient-centred care objectives: results from a qualitative study. BMC Health Serv Res. 2013 Apr 29;13:155. doi: 10.1186/1472-6963-13-155. PMID 23627609
- [Background] MacCarthy D, Kallstrom L, Kadlec H, Hollander M. Improving primary care in British Columbia, Canada: evaluation of a peer-to-peer continuing education program for family physicians. BMC Med Educ. 2012 Nov 9;12:110. doi: 10.1186/1472-6920-12-110. PMID 23140230
- [Background] Pradhan AD, Rifai N, Buring JE, Ridker PM. Hemoglobin A1c predicts diabetes but not cardiovascular disease in nondiabetic women. Am J Med. 2007 Aug;120(8):720-7. doi: 10.1016/j.amjmed.2007.03.022. PMID 17679132
- [Background] Khaw KT, Wareham N, Bingham S, Luben R, Welch A, Day N. Association of hemoglobin A1c with cardiovascular disease and mortality in adults: the European prospective investigation into cancer in Norfolk. Ann Intern Med. 2004 Sep 21;141(6):413-20. doi: 10.7326/0003-4819-141-6-200409210-00006. PMID 15381514
- [Background] Kodama S, Horikawa C, Fujihara K, Hirasawa R, Yachi Y, Yoshizawa S, Tanaka S, Sone Y, Shimano H, Iida KT, Saito K, Sone H. Use of high-normal levels of haemoglobin A(1C) and fasting plasma glucose for diabetes screening and for prediction: a meta-analysis. Diabetes Metab Res Rev. 2013 Nov;29(8):680-92. doi: 10.1002/dmrr.2445. PMID 23963843
- [Background] Bonora E, Tuomilehto J. The pros and cons of diagnosing diabetes with A1C. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S184-90. doi: 10.2337/dc11-s216. No abstract available. PMID 21525453
- [Background] Schwarzer R. Modeling health behavior change: how to predict and modify the adoption and maintenance of health behaviors. Applied Psychology 2008;57(1):1-29
- [Background] Petrella RJ, Aizawa K, Shoemaker K, Overend T, Piche L, Marin M, Shapiro S, Atkin S. Efficacy of a family practice-based lifestyle intervention program to increase physical activity and reduce clinical and physiological markers of vascular health in patients with high normal blood pressure and/or high normal blood glucose (SNAC): study protocol for a randomized controlled trial. Trials. 2011 Feb 16;12:45. doi: 10.1186/1745-6215-12-45. PMID 21324150
- [Background] Petrella RJ, Lattanzio CN. Does counseling help patients get active? Systematic review of the literature. Can Fam Physician. 2002 Jan;48:72-80. PMID 11852615
- [Background] Petrella RJ, Lattanzio CN, Overend TJ. Physical activity counseling and prescription among canadian primary care physicians. Arch Intern Med. 2007 Sep 10;167(16):1774-81. doi: 10.1001/archinte.167.16.1774. PMID 17846397
- [Background] Williford HN, Barfield BR, Lazenby RB, Olson MS. A survey of physicians' attitudes and practices related to exercise promotion. Prev Med. 1992 Sep;21(5):630-6. doi: 10.1016/0091-7435(92)90070-x. PMID 1438111
- [Background] Liu-Ambrose TY, Khan KM, Eng JJ, Gillies GL, Lord SR, McKay HA. The beneficial effects of group-based exercises on fall risk profile and physical activity persist 1 year postintervention in older women with low bone mass: follow-up after withdrawal of exercise. J Am Geriatr Soc. 2005 Oct;53(10):1767-73. doi: 10.1111/j.1532-5415.2005.53525.x. PMID 16181178
- [Background] Davis JC, Marra CA, Beattie BL, Robertson MC, Najafzadeh M, Graf P, Nagamatsu LS, Liu-Ambrose T. Sustained cognitive and economic benefits of resistance training among community-dwelling senior women: a 1-year follow-up study of the Brain Power study. Arch Intern Med. 2010 Dec 13;170(22):2036-8. doi: 10.1001/archinternmed.2010.462. No abstract available. PMID 21149764
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Reliability and validity of a diabetes quality-of-life measure for the diabetes control and complications trial (DCCT). The DCCT Research Group. Diabetes Care. 1988 Oct;11(9):725-32. doi: 10.2337/diacare.11.9.725. PMID 3066604
- [Background] Dolan P, Roberts J. Modelling valuations for Eq-5d health states: an alternative model using differences in valuations. Med Care. 2002 May;40(5):442-6. doi: 10.1097/00005650-200205000-00009. PMID 11961478
- [Background] Davis JC, Liu-Ambrose T, Khan KM, Robertson MC, Marra CA. SF-6D and EQ-5D result in widely divergent incremental cost-effectiveness ratios in a clinical trial of older women: implications for health policy decisions. Osteoporos Int. 2012 Jul;23(7):1849-57. doi: 10.1007/s00198-011-1770-3. Epub 2011 Sep 10. PMID 21909728
- [Background] Davis JC, Marra CA, Robertson MC, Khan KM, Najafzadeh M, Ashe MC, Liu-Ambrose T. Economic evaluation of dose-response resistance training in older women: a cost-effectiveness and cost-utility analysis. Osteoporos Int. 2011 May;22(5):1355-66. doi: 10.1007/s00198-010-1356-5. Epub 2010 Aug 4. PMID 20683707
- [Background] Koopman JJ, van Bodegom D, Jukema JW, Westendorp RG. Risk of cardiovascular disease in a traditional African population with a high infectious load: a population-based study. PLoS One. 2012;7(10):e46855. doi: 10.1371/journal.pone.0046855. Epub 2012 Oct 11. PMID 23071653
- [Background] Hologic Inc. Hologic QDR User's Guide. Bedford, MA: Hologic Inc
- [Background] Anderson TJ, Gregoire J, Hegele RA, Couture P, Mancini GB, McPherson R, Francis GA, Poirier P, Lau DC, Grover S, Genest J Jr, Carpentier AC, Dufour R, Gupta M, Ward R, Leiter LA, Lonn E, Ng DS, Pearson GJ, Yates GM, Stone JA, Ur E. 2012 update of the Canadian Cardiovascular Society guidelines for the diagnosis and treatment of dyslipidemia for the prevention of cardiovascular disease in the adult. Can J Cardiol. 2013 Feb;29(2):151-67. doi: 10.1016/j.cjca.2012.11.032. PMID 23351925
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926
- [Background] Washburn RA, McAuley E, Katula J, Mihalko SL, Boileau RA. The physical activity scale for the elderly (PASE): evidence for validity. J Clin Epidemiol. 1999 Jul;52(7):643-51. doi: 10.1016/s0895-4356(99)00049-9. PMID 10391658
- [Background] Hoppmann CA, Coats AH, Blanchard-Fields F. Goals and everyday problem solving: examining the link between age-related goals and problem-solving strategy use. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2008 Jul;15(4):401-23. doi: 10.1080/13825580701533777. PMID 17899456
- [Background] Slade L, C. H. Time-sampling research in Health Psychology: Potential contributions and new trends. European Health Psychologist 2011;13:65-9
- [Background] Hoppmann C, Gerstorf D. Spousal goals, affect quality, and collaborative problem solving: Evidence from a time-sampling study with older couples. Research in Human Development 2013;10:70-87
- [Background] Drummond MF, Sculpher MJ, Torrance GW, et al. Methods for the Economic Evaluation of Health Care Programmes (Third Edition). New York: Oxford University Press 2005.
- [Background] Davis JC, Robertson MC, Ashe MC, Liu-Ambrose T, Khan KM, Marra CA. Does a home-based strength and balance programme in people aged > or =80 years provide the best value for money to prevent falls? A systematic review of economic evaluations of falls prevention interventions. Br J Sports Med. 2010 Feb;44(2):80-9. doi: 10.1136/bjsm.2008.060988. PMID 20154094
- [Background] Davis JC, Robertson MC, Ashe MC, Liu-Ambrose T, Khan KM, Marra CA. International comparison of cost of falls in older adults living in the community: a systematic review. Osteoporos Int. 2010 Aug;21(8):1295-306. doi: 10.1007/s00198-009-1162-0. Epub 2010 Feb 27. PMID 20195846
- [Background] Marra CA, Cibere J, Grubisic M, Grindrod KA, Gastonguay L, Thomas JM, Embley P, Colley L, Tsuyuki RT, Khan KM, Esdaile JM. Pharmacist-initiated intervention trial in osteoarthritis: a multidisciplinary intervention for knee osteoarthritis. Arthritis Care Res (Hoboken). 2012 Dec;64(12):1837-45. doi: 10.1002/acr.21763. PMID 22930542
- [Background] Woolcott JC, Khan KM, Mitrovic S, Anis AH, Marra CA. The cost of fall related presentations to the ED: a prospective, in-person, patient-tracking analysis of health resource utilization. Osteoporos Int. 2012 May;23(5):1513-9. doi: 10.1007/s00198-011-1764-1. Epub 2011 Sep 3. PMID 21892675
- [Background] Woolcott JC, Richardson KJ, Wiens MO, Patel B, Marin J, Khan KM, Marra CA. Meta-analysis of the impact of 9 medication classes on falls in elderly persons. Arch Intern Med. 2009 Nov 23;169(21):1952-60. doi: 10.1001/archinternmed.2009.357. PMID 19933955
- [Background] Guimaraes C, Marra CA, Colley L, Gill S, Simpson S, Meneilly G, Queiroz RH, Lynd LD. Socioeconomic differences in preferences and willingness-to-pay for insulin delivery systems in type 1 and type 2 diabetes. Diabetes Technol Ther. 2009 Sep;11(9):567-73. doi: 10.1089/dia.2009.0034. PMID 19764835
- [Background] Guimaraes C, Marra CA, Colley L, Gill S, Simpson SH, Meneilly GS, Queiroz RH, Lynd LD. A valuation of patients' willingness-to-pay for insulin delivery in diabetes. Int J Technol Assess Health Care. 2009 Jul;25(3):359-66. doi: 10.1017/S0266462309990055. PMID 19619355
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Derived] Sims Gould J, Tong C, Ly J, Vazirian S, Windt A, Khan K. Process evaluation of team-based care in people aged >65 years with type 2 diabetes mellitus. BMJ Open. 2019 Aug 2;9(8):e029965. doi: 10.1136/bmjopen-2019-029965. PMID 31377711
- [Derived] Khan KM, Windt A, Davis JC, Dawes M, Liu-Ambrose T, Madden K, Marra CA, Housden L, Hoppmann C, Adams DJ. Group Medical Visits (GMVs) in primary care: an RCT of group-based versus individual appointments to reduce HbA1c in older people. BMJ Open. 2015 Jul 13;5(7):e007441. doi: 10.1136/bmjopen-2014-007441. PMID 26169803